CLINICAL TRIAL: NCT06310993
Title: Exercise to Boost Immunity in Advanced Cancer: Feasibility of Combined Aerobic Exercise and Resistance Training for Patients with Advanced Mesothelioma and Pancreatic Cancer
Brief Title: Exercise to Boost Immunity in Advanced Cancer
Acronym: BICEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Sheffield Hallam University (Other); University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH22549
Record Dates: First submitted 2024-02-28; First posted 2024-03-15 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Mesothelioma; Lung; Pancreatic Cancer
MeSH Terms: conditions — Mesothelioma; Pancreatic Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): The exercise programme will include one weekly supervised exercise sessions and one weekly unsupervised exercise session. The frequency will be twice weekly, one supervised and one unsupervised session a week for 12 weeks. The exercises will be of moderate intensity aerobic interval exercise (performing at 60% maximum heart rate) combined with 1-3 sets of 6-12 Repetition Maximum (RM) resistance training. The type of exercise will be aerobic interval exercise (cycling) and Resistance training (3 exercises: chest press, biceps, and leg curl) The timing will be 4 x 4-minute cycling at 60%, max HR with 3 minutes active recovery. 3 sets with 2 minutes per set - around 20 minutes resistance training
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise programme is the intervention for this study

SUMMARY:
The trial is a prospective feasibility trial conducted in Sheffield. Recruitment will include twenty patients receiving first line palliative immunotherapy for advanced, unresectable or metastatic mesothelioma and patients receiving first line systemic anti-cancer treatment for pancreatic cancer. Patients will attend the AWRC for a supervised exercise session once a week to include aerobic exercise along with an unsupervised weekly exercise session for 3 months. Blood samples will be collected at baseline and then monthly for 3 months, pre and post the supervised exercise session. Cytokine, myokine and immune cell concentration will be analysed using cytokine bead-based multiplex immune assays and RNA-seq to full profile changes in gene and protein expression

DETAILED DESCRIPTION:
Immunotherapy is rapidly revolutionising cancer care with ICIs demonstrating clinical efficacy in multiple cancer settings and are indicated in the peri-operative, advanced, and recurrent settings for various tumour types. Mesothelioma is classed as a "hot tumour" due to its lymphocyte rich tumour microenvironment which has demonstrated some clinical response to immunotherapy. On the other end of the spectrum, 'cold tumours' such as pancreatic cancer, have been shown to have low immune cell populations and reduced immune activity within their tumour microenvironments. Evidence suggests that in cancer patients, exercise improves overall health, may prolong survival as well as reduce cancer-related fatigue and modulate the immune system through multiple mechanisms. Physical activity is defined as 'any bodily movement produced by skeletal muscles or that requires contraction of your muscles and energy expenditure. Exercise-induced leucocytosis refers to the immediate increase in circulatory leukocytes after a single exercise activity. The use of exercise as medicine requires an understanding of the appropriate dose which is highly dependent on the FITT principles (Frequency, Intensity, Time, and Type) and this is crucial for generating desired outcomes. Although ICIs have revolutionised treatment for many different cancers, less than 40% of patients derive significant benefit from ICIs which highlights the need to improve responsiveness The primary objective is to determine the feasibility of exercise during systemic anti-cancer treatment in patients with advanced mesothelioma or pancreatic cancer.

The secondary objectives are:

iTo determine the safety of exercise during systemic anti-cancer treatment in patients with advanced mesothelioma or pancreatic cancer.

ii. To determine the acceptability of exercise during systemic anti-cancer treatment in patients with advanced mesothelioma or pancreatic cancer.

iii. Does exercise boost immune cell activation in cancer patients? iv. To determine the effect of exercise on cytokine/ myokine levels in the blood v.To determine the effect of exercise on radiological response or progression. vi.To determine the effect of exercise on lung function.

ELIGIBILITY:
Inclusion Criteria:

* Patients about to start or who are undergoing first line palliative immunotherapy for advanced, unresectable, or metastatic mesothelioma or patients about to start or who are undergoing first line palliative chemotherapy for advanced, unresectable, or metastatic pancreatic cancer.
* Age over 18 years old
* Histological or cytological diagnosis of mesothelioma or pancreatic cancer.
* ECOG Performance status 0-1 (to be assessed by clinician)
* Ability to provide informed consent

Exclusion Criteria:

* Prior treatment with systemic anti-cancer treatment
* More than one primary cancer
* Uncontrolled brain or bone metastases
* Patients who have progressed on first line palliative immunotherapy for advanced, unresectable, or metastatic mesothelioma.
* Patients who have progressed on first line palliative chemotherapy for advanced, unresectable, or metastatic pancreatic cancer.
* Patients with active co-morbidities that would prevent or limit their participation in the exercise intervention
* Age below 18 years old
* No histological or cytological diagnosis of mesothelioma or pancreatic cancer.
* ECOG Performance status of 2 or more
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | completion of the 12-week exercise intervention
  Adherence rate: The ratio of the number of exercise sessions performed to the number of exercise sessions planned.

SECONDARY OUTCOMES:
Secondary outcome 1 | completion of the 12-week exercise intervention
  The number of directly related adverse events.
Secondary Outcome 2 | completion of the 12-week exercise intervention
  Acceptability rate: the ratio of those recruited to the trial to those approached as eligible.
Secondary Outcome 3 | completion of the 12-week exercise intervention
  Attrition rate: the ratio of dropouts from the trial to those enrolled initially.
Secondary Outcome 4 | Baseline, then 4-weekly pre- and post- exercise interventions for 12 weeks and then at completion of the 12-week exercise intervention
  Peripheral blood mononuclear cells (PBMC) in the blood. Immune cell activation will be determined by an increased in cytotoxic immune components (Natural Killer cells / CD8 T cells) and a decrease in immunosuppressive immune cells (regulatory T cells).
Secondary Outcome 5 | Baseline, then 4-weekly pre- and post- exercise interventions for 12 weeks and then at completion of the 12-week exercise intervention.
  The levels of cytokines/ myokines in the blood
Secondary Outcome 6 | Baseline and at 12 weeks
  Evidence of radiological response or progression as per RECIST 1.1 reporting of CT scans
Secondary Outcome 7 | Baseline and at 12 weeks
  Lung function as per results of lung function tests

CONTACTS AND LOCATIONS:
Overall Officials: Brindley Hapuarachi, MD, Principal Investigator — Sheffield Teaching Hospitals NHS FT
Locations (2):
- United Kingdom (2):
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Sheffield Hallam University, Sheffield, South Yorkshire

IPD SHARING:
Plan to Share IPD: No